CLINICAL TRIAL: NCT03022513
Title: Fibromyalgia-like Joint/Muscle Pain and Synovitis in Non-celiac Wheat Sensitivity Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ACPM13
Record Dates: First submitted 2016-12-30; First posted 2017-01-16 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Non-celiac Wheat Sensitivity
Keywords: Non-celiac Wheat Sensitivity; fibromyalgia; synovitis
MeSH Terms: conditions — Fibromyalgia; Synovitis | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NCWS patients (Active Comparator): Fifty consecutive adult patients with an irritable bowel syndrome (IBS)-like clinical presentation, according to Rome III criteria, and a definitive diagnosis of NCWS. The patients will be recruited between January 2017 and January 2018 at 2 centers: the Department of Internal Medicine at the University Hospital of Palermo, Italy, and the Department of Internal Medicine of the Hospital of Sciacca, Agrigento, Italy. All subjects will undergo clinical evaluation and hands and feet joints ultrasonography at the Rheumatology Unit of the University of Palermo, Italy.
  Interventions: Other: Gluten free diet
- CD patients (No Intervention): Fifty sex- and age-matched subjects with CD, diagnosed according to standard criteria during the same study period and enrolled, at the same 2 centers, as first control group. All subjects will undergo clinical evaluation and hands and feet joints ultrasonography at the Rheumatology Unit of the University of Palermo, Italy.
- IBS patients (No Intervention): Fifty sex- and age-matched subjects with IBS unrelated to NCWS or other food 'intolerance', diagnosed according to standard criteria during the same study period and enrolled, at the same 2 centers, as second control group. All subjects will undergo clinical evaluation and hands and feet joints ultrasonography at the Rheumatology Unit of the University of Palermo.

INTERVENTIONS:
Other: Gluten free diet — The investigators will evaluate the prevalence of fibromyalgia-like joint/muscle pain and the possible ultrasonographical alterations (i.e. synovitis) of hands and feet joints in NCWS patient at baseline (i.e. at the moment of diagnosis) and after a gluten free diet period of almost 6 months.
  Arms: NCWS patients

SUMMARY:
Recently it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal and/or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). Nowadays no data are available on the characteristic of 'rheumatologic' symptoms of NCWS patients. Therefore, the aims of the present study are: 1) to investigate the prevalence of fibromyalgia-like joint/muscle pain in NCWS patient, 2) to search for possible ultrasonographic alterations (i.e. synovitis) of hands and feet joints of NCWS patients, and 3) to evaluate modification of fibromyalgia-like joint/muscle pain in NCWS patients after a gluten free diet period of almost 6 months.

DETAILED DESCRIPTION:
Recently it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. CD is an immunological disorder whose best-known manifestations are gastrointestinal symptoms. However, early joint manifestations are common and frequently overlooked features of the disease. Similarly, the clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal and/or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). Nowadays no data are available on the characteristic of 'rheumatological' symptoms of NCWS patients. Therefore, the aims of the present study are: 1) to investigate the prevalence of fibromyalgia-like joint/muscle pain in NCWS patient, 2) to search for possible ultrasonographical alterations (i.e. synovitis) of hands and feet joints of NCWS patients, and 3) to evaluate modification of fibromyalgia-like joint/muscle pain in NCWS patients after a gluten free diet period of almost 6 months.

ELIGIBILITY:
Inclusion Criteria:

All the patients met the recently proposed criteria:

* negative serum anti-tissue transglutaminase and antiendomysium (EmA) immunoglobulin (Ig) A and IgG antibodies
* absence of intestinal villous atrophy
* IgE-mediated immunoallergic tests negative to wheat and cow's milk protein (skin prick tests and/or serum specific IgE detection).

Adjunctive criteria adopted in our patients were:

* resolution of the gastrointestinal and extra-intestinal symptoms on a standard elimination diet, without wheat, cow's milk, egg, tomato, chocolate, or other food(s) causing self-reported symptoms
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge, performed as described previously. DBPC cow's milk protein challenge will be also performed to diagnose cow's milk protein allergy.

Exclusion Criteria:

Exclusion criteria will be:

* age <18 years
* positive EmA in the culture medium of the duodenal biopsies, even if the villi to crypts ratio in the duodenal mucosa was normal
* self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study
* other organic gastrointestinal diseases
* previously diagnosed rheumatic diseases
* nervous system disease and/or major psychiatric disorder
* physical impairment limiting physical activity
* menopause; steroid and sex steroid therapy, hormone replacement therapy or ovariectomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of fibromyalgia-like joint/muscle pain in NCWS patients | up to 12 months
  Prevalence of fibromyalgia-like joint/muscle pain in NCWS patient using an ad hoc questionnaire and orientated clinical examination (tenders and triggers point evaluation)
Hands and feet joints ultrasonography alterations | up to 12 months
  Hands and feet joints ultrasonography alterations in NCWS patients.

SECONDARY OUTCOMES:
Modification of fibromyalgia-like joint/muscle pain in NCWS patients after gluten free diet | up to 12 months
  Modification of fibromyalgia-like joint/muscle pain, by visual analogic scale, in NCWS patients after a gluten free diet period of almost 6 months.
Modifications of hands and feet joints ultrasonography alterations in NCWS patients after gluten free diet | up to 12 months
  Modifications of hands and feet joints ultrasonography alterations in NCWS patients after a gluten free diet period of almost 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210